CLINICAL TRIAL: NCT02774265
Title: A Different Approach to Preventing Thrombosis (ADAPT): A Randomized Controlled Trial Comparing Low Molecular Weight Heparin to Acetylsalicylic Acid in Orthopedic Trauma Patients
Brief Title: A Different Approach to Preventing Thrombosis
Acronym: ADAPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Deborah Stein, Professor of Surgery, Chief of Trauma, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00065750
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Venous Thromboembolism; Pulmonary Embolism
Keywords: Fracture; Prophylaxis
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Fractures, Bone | interventions — Enoxaparin; BID protein, human; Heparin, Low-Molecular-Weight; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VTE prophylaxis with Enoxaparin 30mg BID (Active Comparator): The group receiving VTE prophylaxis with enoxaparin 30mg subcutaneous BID.
  Interventions: Drug: VTE prophylaxis with Enoxaparin 30mg BID
- VTE prophylaxis with Aspirin 81mg BID (Active Comparator): The group receiving VTE prophylaxis with ASA 81mg PO BID
  Interventions: Drug: VTE prophylaxis with Aspirin 81mg BID

INTERVENTIONS:
Drug: VTE prophylaxis with Enoxaparin 30mg BID — Patients will receive Enoxaparin 30mg BID for DVT prophylaxis and will be followed to determine the efficacy, safety and cost when used for VTE prophylaxis in high-risk orthopedic traumas administered for the length of time indicated by standard of care based on the injury.
  Other Names: Lovenox; Low Molecular Weight Heparin (LMWH)
  Arms: VTE prophylaxis with Enoxaparin 30mg BID
Drug: VTE prophylaxis with Aspirin 81mg BID — Patients will receive Aspirin 81mg BID for DVT prophylaxis and will be followed to determine the efficacy, safety and cost when used for VTE prophylaxis in high-risk orthopedic traumas administered for the length of time indicated by standard of care based on the injury.
  Other Names: ASA (Acetylsalicylic Acid)
  Arms: VTE prophylaxis with Aspirin 81mg BID

SUMMARY:
The purpose of this study is to perform a pragmatic randomized controlled trial to compare the use of low molecular weight heparin (LMWH, lovenox, enoxaparin) versus acetylsalicylic acid (ASA) for venous thromboembolism (VTE) prophylaxis in patients with high-risk lower extremity fractures.

DETAILED DESCRIPTION:
Purpose:

To perform a pragmatic randomized controlled trial of the use of low molecular weight heparin (LMWH, enoxaparin, lovenox) versus Aspirin (ASA) for VTE prophylaxis in patients with high-risk extremity fractures.

Specific Aims:

1. To compare the bleeding complication outcomes associated with LMWH versus ASA in patients receiving VTE prophylaxis following high-risk lower extremity fractures.
2. To compare the incidence of clinically important VTE events associated with LMWH versus ASA for VTE prophylaxis in patients receiving VTE prophylaxis following high-risk lower extremity fractures.
3. To compare the 6-month treatment costs associated with VTE prophylaxis using either LMWH or ASA for high-risk lower extremity fracture patients

Hypothesis:

1. Among patients with high risk lower extremity fractures receiving VTE prophylaxis, the rate of bleeding complications will be lower for patients receiving ASA compared to those receiving LMWH.
2. Among patients with high risk lower extremity fractures receiving VTE prophylaxis, the rate of VTE for patients receiving ASA will be no greater than those receiving LMWH.
3. Among patients with high risk lower extremity fractures receiving VTE prophylaxis, the 6-month treatment costs will be lower for patients receiving ASA compared to those receiving LMWH.

Methods/Outcomes:

A randomized controlled trial will be conducted to assess the use of LMWH versus ASA for VTE prophylaxis in patients with high-risk extremity fractures.

The aim-specific outcomes to be collected are as follows:

1. A composite of the following major bleeding related complications:

   1. Fatal bleeding into a critical organ (retroperitoneal, intracranial, intraocular, intraspinal)
   2. Clinically overt bleed with a > 2g/dL drop in Hb or requiring > 2U transfusion
   3. Wound drainage or hematoma requiring reoperation
   4. Diagnosis of deep surgical site infection
2. VTE Events defined as a composite of any symptomatic proximal DVT (in the femoral or popliteal vessels), or PE (central, segmental or subsegmental). All VTE events will be confirmed using multiplanar CT scan or formal venous duplex exam.
3. Cost of VTE prophylaxis treatment, VTE events and bleeding related complications.

Data Collection:

Patients meeting inclusion/exclusion criteria will be prospectively randomized to one of two treatment arms. Block randomization will be used. Patients will receive VTE prophylaxis as allocated, and followed for their index hospitalization and a 3month period post discharge for VTE events and bleeding complications. Outcome data will be prospectively collected during index hospitalization, and at 2 weeks and 3 months post discharge, and blind analysis and interpretation of results will be performed at 50% and 100% recruitment.

Data Analysis:

All data will be reported as mean and standard deviations for continuous variables and proportions and percentages for categorical data. Kaplan-Meier survival and Cox proportional hazard analysis will be completed for time to VTE and bleeding complication outcomes. Sub-group analysis will include Injury Severity Score and fracture location. An independent Data Safety and Monitoring Committee will complete interim analysis at 50% recruitment. A cost analysis will be conducted using a 6month and lifetime time horizon with a societal perspective. Component costs will consist of: VTE prophylaxis costs, unscheduled follow-ups, emergency room visit, hospital admission or unscheduled repeat surgical intervention for VTE or bleeding complications.

Study Treatment Arms:

1. VTE prophylaxis with Enoxaparin 30mg SC BID
2. VTE prophylaxis with ASA 81mg PO BID

ELIGIBILITY:
Inclusion Criteria:

* All patients treated at a level-1 trauma center with any one or more of the following injuries: Pelvis fracture (operative or non-operative), Acetabulum fracture (operative or non-operative), or any operative extremity fracture (proximal to metatarsals/carpals)
* Age greater than or equal to 18 years old

Exclusion Criteria:

* Patients receiving pre-existing confounding prophylaxis or therapeutic anticoagulation (not to include anti-platelet agents) prior to admission or those receiving greater than one dose of LMWH since injury
* Patients with pre-existing coagulopathy
* Patients with a previous history of VTE within the last 6 months
* Patients who are pregnant
* Patients with CNS or spinal cord injury with potential need for further neurosurgical intervention precluding anticoagulation with aspirin
* Patients with active bleeding precluding the use of anticoagulation
* Impaired creatinine clearance <30ml/min at the time of randomization
* History of Heparin Induced Thrombocytopenia or ASA or NSAID allergy
* Prisoners
* Non-english speaking patients
* Patients who have an indication for therapeutic anticoagulation
* Patients deemed inappropriate for inclusion in the study by their treating physician. Reason must be documented
* Patients who would not normally receive VTE prophylaxis for their injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Stein, MD, MPH, Principal Investigator — R. Adams Cowley Shock Trauma Center
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared as aggregate data only to protect the identity of individual participants.

REFERENCES:
- [Background] Cohen AT, Imfeld S, Markham J, Granziera S. The use of aspirin for primary and secondary prevention in venous thromboembolism and other cardiovascular disorders. Thromb Res. 2015 Feb;135(2):217-25. doi: 10.1016/j.thromres.2014.11.036. Epub 2014 Dec 13. PMID 25541030
- [Background] Selby R, Geerts WH, Kreder HJ, Crowther MA, Kaus L, Sealey F; D-KAF (Dalteparin in Knee-to-Ankle Fracture) Investigators. A double-blind, randomized controlled trial of the prevention of clinically important venous thromboembolism after isolated lower leg fractures. J Orthop Trauma. 2015 May;29(5):224-30. doi: 10.1097/BOT.0000000000000250. PMID 25900749
- [Background] Scolaro JA, Taylor RM, Wigner NA. Venous thromboembolism in orthopaedic trauma. J Am Acad Orthop Surg. 2015 Jan;23(1):1-6. doi: 10.5435/JAAOS-23-01-1. PMID 25538125
- [Background] Gritsiouk Y, Hegsted DA, Schlesinger P, Gardiner SK, Gubler KD. A retrospective analysis of the effectiveness of low molecular weight heparin for venous thromboembolism prophylaxis in trauma patients. Am J Surg. 2014 May;207(5):648-51; discussion 651-2. doi: 10.1016/j.amjsurg.2013.12.010. Epub 2014 Jan 30. PMID 24560359
- [Background] Schousboe JT, Brown GA. Cost-effectiveness of low-molecular-weight heparin compared with aspirin for prophylaxis against venous thromboembolism after total joint arthroplasty. J Bone Joint Surg Am. 2013 Jul 17;95(14):1256-64. doi: 10.2106/JBJS.L.00400. PMID 23864173
- [Background] Lieberman JR, Pensak MJ. Prevention of venous thromboembolic disease after total hip and knee arthroplasty. J Bone Joint Surg Am. 2013 Oct 2;95(19):1801-11. doi: 10.2106/JBJS.L.01328. PMID 24088973
- [Background] Mortazavi SM, Hansen P, Zmistowski B, Kane PW, Restrepo C, Parvizi J. Hematoma following primary total hip arthroplasty: a grave complication. J Arthroplasty. 2013 Mar;28(3):498-503. doi: 10.1016/j.arth.2012.07.033. Epub 2012 Oct 31. PMID 23122656
- [Background] Brakenridge SC, Henley SS, Kashner TM, Golden RM, Paik DH, Phelan HA, Cohen MJ, Sperry JL, Moore EE, Minei JP, Maier RV, Cuschieri J; Inflammation and the Host Response to Injury Investigators. Comparing clinical predictors of deep venous thrombosis versus pulmonary embolus after severe injury: a new paradigm for posttraumatic venous thromboembolism? J Trauma Acute Care Surg. 2013 May;74(5):1231-7; discussion 1237-8. doi: 10.1097/TA.0b013e31828cc9a0. PMID 23609272
- [Background] Sagi HC, Dziadosz D, Mir H, Virani N, Olson C. Obesity, leukocytosis, embolization, and injury severity increase the risk for deep postoperative wound infection after pelvic and acetabular surgery. J Orthop Trauma. 2013 Jan;27(1):6-10. doi: 10.1097/BOT.0b013e31825cf382. PMID 23263468
- [Background] Raphael IJ, Tischler EH, Huang R, Rothman RH, Hozack WJ, Parvizi J. Aspirin: an alternative for pulmonary embolism prophylaxis after arthroplasty? Clin Orthop Relat Res. 2014 Feb;472(2):482-8. doi: 10.1007/s11999-013-3135-z. PMID 23817755
- [Background] Stewart DW, Freshour JE. Aspirin for the prophylaxis of venous thromboembolic events in orthopedic surgery patients: a comparison of the AAOS and ACCP guidelines with review of the evidence. Ann Pharmacother. 2013 Jan;47(1):63-74. doi: 10.1345/aph.1R331. Epub 2013 Jan 16. PMID 23324504
- [Background] Anderson DR, Dunbar MJ, Bohm ER, Belzile E, Kahn SR, Zukor D, Fisher W, Gofton W, Gross P, Pelet S, Crowther M, MacDonald S, Kim P, Pleasance S, Davis N, Andreou P, Wells P, Kovacs M, Rodger MA, Ramsay T, Carrier M, Vendittoli PA. Aspirin versus low-molecular-weight heparin for extended venous thromboembolism prophylaxis after total hip arthroplasty: a randomized trial. Ann Intern Med. 2013 Jun 4;158(11):800-6. doi: 10.7326/0003-4819-158-11-201306040-00004. PMID 23732713
- [Background] Cossetto DJ, Goudar A, Parkinson K. Safety of peri-operative low-dose aspirin as a part of multimodal venous thromboembolic prophylaxis for total knee and hip arthroplasty. J Orthop Surg (Hong Kong). 2012 Dec;20(3):341-3. doi: 10.1177/230949901202000315. PMID 23255642
- [Background] Vulcano E, Gesell M, Esposito A, Ma Y, Memtsoudis SG, Gonzalez Della Valle A. Aspirin for elective hip and knee arthroplasty: a multimodal thromboprophylaxis protocol. Int Orthop. 2012 Oct;36(10):1995-2002. doi: 10.1007/s00264-012-1588-4. Epub 2012 Jun 12. PMID 22684546
- [Background] Mont MA, Jacobs JJ. AAOS clinical practice guideline: preventing venous thromboembolic disease in patients undergoing elective hip and knee arthroplasty. J Am Acad Orthop Surg. 2011 Dec;19(12):777-8. doi: 10.5435/00124635-201112000-00008. No abstract available. PMID 22134210
- [Background] Bozic KJ, Vail TP, Pekow PS, Maselli JH, Lindenauer PK, Auerbach AD. Does aspirin have a role in venous thromboembolism prophylaxis in total knee arthroplasty patients? J Arthroplasty. 2010 Oct;25(7):1053-60. doi: 10.1016/j.arth.2009.06.021. Epub 2009 Aug 12. PMID 19679434
- [Background] Hill J, Treasure T; Guideline Development Group. Reducing the risk of venous thromboembolism (deep vein thrombosis and pulmonary embolism) in patients admitted to hospital: summary of the NICE guideline. Heart. 2010 Jun;96(11):879-82. doi: 10.1136/hrt.2010.198275. No abstract available. PMID 20478866
- [Background] Slobogean GP, Lefaivre KA, Nicolaou S, O'Brien PJ. A systematic review of thromboprophylaxis for pelvic and acetabular fractures. J Orthop Trauma. 2009 May-Jun;23(5):379-84. doi: 10.1097/BOT.0b013e3181a5369c. PMID 19390367
- [Background] Goel DP, Buckley R, deVries G, Abelseth G, Ni A, Gray R. Prophylaxis of deep-vein thrombosis in fractures below the knee: a prospective randomised controlled trial. J Bone Joint Surg Br. 2009 Mar;91(3):388-94. doi: 10.1302/0301-620X.91B3.20820. PMID 19258618
- [Background] Novicoff WM, Brown TE, Cui Q, Mihalko WM, Slone HS, Saleh KJ. Mandated venous thromboembolism prophylaxis: possible adverse outcomes. J Arthroplasty. 2008 Sep;23(6 Suppl 1):15-9. doi: 10.1016/j.arth.2008.04.014. Epub 2008 Jun 13. PMID 18555656
- [Background] Watson HG, Chee YL. Aspirin and other antiplatelet drugs in the prevention of venous thromboembolism. Blood Rev. 2008 Mar;22(2):107-16. doi: 10.1016/j.blre.2007.11.001. Epub 2008 Jan 15. PMID 18226435
- [Background] Myers DD Jr, Wrobleski SK, Longo C, Bedard PW, Kaila N, Shaw GD, Londy FJ, Rohrer SE, Fex BA, Zajkowski PJ, Meier TR, Hawley AE, Farris DM, Ballard NE, Henke PK, Schaub RG, Wakefield TW. Resolution of venous thrombosis using a novel oral small-molecule inhibitor of P-selectin (PSI-697) without anticoagulation. Thromb Haemost. 2007 Mar;97(3):400-7. PMID 17334507
- [Background] Slavik RS, Chan E, Gorman SK, de Lemos J, Chittock D, Simons RK, Wing PC, Ho SG. Dalteparin versus enoxaparin for venous thromboembolism prophylaxis in acute spinal cord injury and major orthopedic trauma patients: 'DETECT' trial. J Trauma. 2007 May;62(5):1075-81; discussion 1081. doi: 10.1097/TA.0b013e31804fa177. PMID 17495705
- [Background] Burnett RS, Clohisy JC, Wright RW, McDonald DJ, Shively RA, Givens SA, Barrack RL. Failure of the American College of Chest Physicians-1A protocol for lovenox in clinical outcomes for thromboembolic prophylaxis. J Arthroplasty. 2007 Apr;22(3):317-24. doi: 10.1016/j.arth.2007.01.007. PMID 17400085
- [Background] Stannard JP, Lopez-Ben RR, Volgas DA, Anderson ER, Busbee M, Karr DK, McGwin GR Jr, Alonso JE. Prophylaxis against deep-vein thrombosis following trauma: a prospective, randomized comparison of mechanical and pharmacologic prophylaxis. J Bone Joint Surg Am. 2006 Feb;88(2):261-6. doi: 10.2106/JBJS.D.02932. PMID 16452735
- [Background] Myers DD Jr, Rectenwald JE, Bedard PW, Kaila N, Shaw GD, Schaub RG, Farris DM, Hawley AE, Wrobleski SK, Henke PK, Wakefield TW. Decreased venous thrombosis with an oral inhibitor of P selectin. J Vasc Surg. 2005 Aug;42(2):329-36. doi: 10.1016/j.jvs.2005.04.045. PMID 16102635
- [Background] Steele N, Dodenhoff RM, Ward AJ, Morse MH. Thromboprophylaxis in pelvic and acetabular trauma surgery. The role of early treatment with low-molecular-weight heparin. J Bone Joint Surg Br. 2005 Feb;87(2):209-12. doi: 10.1302/0301-620x.87b2.14447. PMID 15736745
- [Background] Jorgensen PS, Warming T, Hansen K, Paltved C, Vibeke Berg H, Jensen R, Kirchhoff-Jensen R, Kjaer L, Kerbouche N, Leth-Espensen P, Narvestad E, Rasmussen SW, Sloth C, Torholm C, Wille-Jorgensen P. Low molecular weight heparin (Innohep) as thromboprophylaxis in outpatients with a plaster cast: a venografic controlled study. Thromb Res. 2002 Mar 15;105(6):477-80. doi: 10.1016/s0049-3848(02)00059-2. PMID 12091045
- [Background] Rogers FB, Cipolle MD, Velmahos G, Rozycki G, Luchette FA. Practice management guidelines for the prevention of venous thromboembolism in trauma patients: the EAST practice management guidelines work group. J Trauma. 2002 Jul;53(1):142-64. doi: 10.1097/00005373-200207000-00032. No abstract available. PMID 12131409
- [Background] Lassen MR, Borris LC, Nakov RL. Use of the low-molecular-weight heparin reviparin to prevent deep-vein thrombosis after leg injury requiring immobilization. N Engl J Med. 2002 Sep 5;347(10):726-30. doi: 10.1056/NEJMoa011327. PMID 12213943
- [Background] Brookenthal KR, Freedman KB, Lotke PA, Fitzgerald RH, Lonner JH. A meta-analysis of thromboembolic prophylaxis in total knee arthroplasty. J Arthroplasty. 2001 Apr;16(3):293-300. doi: 10.1054/arth.2001.21499. PMID 11307125
- [Background] Hak DJ. Prevention of venous thromboembolism in trauma and long bone fractures. Curr Opin Pulm Med. 2001 Sep;7(5):338-43. doi: 10.1097/00063198-200109000-00015. PMID 11584186
- [Background] Prevention of pulmonary embolism and deep vein thrombosis with low dose aspirin: Pulmonary Embolism Prevention (PEP) trial. Lancet. 2000 Apr 15;355(9212):1295-302. PMID 10776741
- [Background] Greenfield LJ, Proctor MC, Rodriguez JL, Luchette FA, Cipolle MD, Cho J. Posttrauma thromboembolism prophylaxis. J Trauma. 1997 Jan;42(1):100-3. doi: 10.1097/00005373-199701000-00017. PMID 9003265
- [Background] Lotke PA, Palevsky H, Keenan AM, Meranze S, Steinberg ME, Ecker ML, Kelley MA. Aspirin and warfarin for thromboembolic disease after total joint arthroplasty. Clin Orthop Relat Res. 1996 Mar;(324):251-8. doi: 10.1097/00003086-199603000-00031. PMID 8595765
- [Background] Collaborative overview of randomised trials of antiplatelet therapy--III: Reduction in venous thrombosis and pulmonary embolism by antiplatelet prophylaxis among surgical and medical patients. Antiplatelet Trialists' Collaboration. BMJ. 1994 Jan 22;308(6923):235-46. PMID 8054013
- [Background] Schumacher WA, Heran CL. Effect of thromboxane receptor antagonists on venous thrombosis in rats. J Pharmacol Exp Ther. 1989 Mar;248(3):1109-15. PMID 2522985
- [Background] Vesterqvist O, Green K, Johnsson H. Thromboxane and prostacyclin formation in patients with deep vein thrombosis. Thromb Res. 1987 Feb 15;45(4):393-402. doi: 10.1016/0049-3848(87)90228-3. PMID 3554598
- [Background] McKenna R, Galante J, Bachmann F, Wallace DL, Kaushal PS, Meredith P. Prevention of venous thromboembolism after total knee replacement by high-dose aspirin or intermittent calf and thigh compression. Br Med J. 1980 Feb 23;280(6213):514-7. doi: 10.1136/bmj.280.6213.514. PMID 6989432
- [Background] Harris WH, Salzman EW, Athanasoulis CA, Waltman AC, DeSanctis RW. Aspirin prophylaxis of venous thromboembolism after total hip replacement. N Engl J Med. 1977 Dec 8;297(23):1246-9. doi: 10.1056/NEJM197712082972302. PMID 335247

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited inpatients admitted between January 19, 2016 and November 1, 2016.
Period: Overall Study
Arm/Group | VTE Prophylaxis With Enoxaparin 30mg BID | VTE Prophylaxis With Aspirin 81mg BID
Started | 164 | 165
Completed | 151 | 159
Not Completed | 13 | 6

BASELINE CHARACTERISTICS:
Population: Analysis is the same as the assignment in Participant Flow
Groups:
- Total: Total of all reporting groups
Arm/Group | VTE Prophylaxis With Enoxaparin 30mg BID | VTE Prophylaxis With Aspirin 81mg BID | Total
Number analyzed (Participants) | 164 | 165 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (20.4) | 48 (18.6) | 46.7 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 61 | 106
  Male | 119 | 104 | 223
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 53 | 45 | 98
  White | 97 | 106 | 203
  More than one race | 6 | 3 | 9
  Unknown or Not Reported | 8 | 11 | 19
Current smoker [Count of Participants; unit: Participants] | 62 | 65 | 127

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Bleeding Events as Assessed by the Need for Blood Transfusions and Procedures for Bleeding Complications After Initiation of the Study Medication.
Description: Includes a greater than 2g/dL drop in hemoglobin, blood transfusion, hematoma evacuation, re-operation for a deep surgical site infection or minor procedure for bleeding and GI bleed
Time Frame: 90 days
Population: As described in Participant Flow
Measure: Count of Participants; unit: Participants
Arm/Group | VTE Prophylaxis With Enoxaparin 30mg BID | VTE Prophylaxis With Aspirin 81mg BID
Number analyzed (Participants) | 164 | 165
Participants | 52 | 53

2. Secondary Outcome: Number of Participants With Deep Venous Thromboembolism
Description: DVT and how the diagnosis was made will be recorded. The number of events in participants in each arm will be compared to evaluate efficacy.
Time Frame: 90 days
Population: same as flow chart
Measure: Count of Participants; unit: Participants
Arm/Group | VTE Prophylaxis With Enoxaparin 30mg BID | VTE Prophylaxis With Aspirin 81mg BID
Number analyzed (Participants) | 164 | 165
Participants | 5 | 9

3. Secondary Outcome: Number of Participants With Pulmonary Embolism Events
Description: Bases on imaging obtained for symptoms.
Time Frame: 90 days
Population: As per flow sheet
Measure: Count of Participants; unit: Participants
Arm/Group | VTE Prophylaxis With Enoxaparin 30mg BID | VTE Prophylaxis With Aspirin 81mg BID
Number analyzed (Participants) | 164 | 165
Participants | 6 | 2

ADVERSE EVENTS:
Time Frame: 90 days post injury
Description: Adverse events as described by our IRB reporting protocol include only unexpected adverse events. Since study outcomes like bleeding and venous thromboembolism are expected, measured outcomes, these are not included.
Arm/Group | VTE Prophylaxis With Enoxaparin 30mg BID | VTE Prophylaxis With Aspirin 81mg BID
All-Cause Mortality (participants affected / at risk) | 3/164 | 3/165
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/165
Other Adverse Events (participants affected / at risk) | 0/164 | 0/165

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT02774265/Prot_SAP_001.pdf